CLINICAL TRIAL: NCT01960166
Title: Impact of Active vs Passive Distraction on Procedural Pain/Distress in the Pediatric Emergency
Brief Title: Active vs Passive Distraction on Procedural Pain in the Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-2254
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Pain Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active distraction (Experimental): Child will use Ipad as active distraction
  Interventions: Behavioral: Active Distraction
- Passive Distraction (Experimental): Child will watch movie as passive distraction (control)
  Interventions: Behavioral: Passive Distraction

INTERVENTIONS:
Behavioral: Active Distraction — iPad will be used as active distraction
  Arms: Active distraction
Behavioral: Passive Distraction — child will watch TV as passive distraction
  Arms: Passive Distraction

SUMMARY:
The investigators proposed study will investigate the efficacy of tablet computer distraction as an analgesic for the pain associated with various painful procedures in the emergency department. Since prior studies have shown that distraction by a parent or nurse can be an effective analgesic, there is reason to believe that tablet computer distraction will similarly reduce pain. Participants in the control group will receive a cartoon on the TV monitor in the patient room, while participants in the study group will receive a more immersive distraction of playing a game or watching a cartoon (for children too young to play a game) on a tablet computer. Data from this study will help inform best practices for administering painful procedures in a way that minimizes pain.

ELIGIBILITY:
Inclusion Criteria:

Healthy pediatric patients in the University of Chicago emergency department who are undergoing insertion of a peripheral intravenous line, intramuscular injection, fingerstick, subcutaneous injection, laceration repair (sutures, tissue adhesive, and staples), nail avulsion, or abscess incision and drainage.

Exclusion Criteria:

Non-English speaking, over the age of 18 trauma, have come in for asthma-related complaints, are being resuscitated, are neurosurgical/neurology/seizure patients, or patients in whom use of distraction would interfere with the procedure

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Score on pain scale | after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Gray, MD, Principal Investigator — University of Chicago
Locations (1):
- U of Chicago Medical Center, Chicago, Illinois, United States